CLINICAL TRIAL: NCT02656667
Title: Effect of Neuromuscular Electrical Stimulation Versus Cycle Ergometer Training in a Pulmonary Rehabilitation Program
Acronym: ESNM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ESNM (RB 15.058)
Record Dates: First submitted 2016-01-06; First posted 2016-01-15 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2019-04

CONDITIONS: COPD
Keywords: COPD pulmonary rehabilitation; neuromuscular electrical stimulation; sit to stand test COPD; quadriceps strengthening
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- neuromuscular electrical stimulation (Experimental): conventional pulmonary rehabilitation including exercise training on treadmill and neuromuscular electrical stimulation with a medical device for quadriceps muscle strengthening
  Interventions: Device: neuromuscular electrical stimulation; Other: Conventional pulmonary rehabilitation
- cycle ergometer training (Experimental): conventional pulmonary rehabilitation including exercise training on treadmill and quadriceps strenghthening on cycle-ergometer
  Interventions: Device: cycle ergometer training; Other: Conventional pulmonary rehabilitation

INTERVENTIONS:
Device: neuromuscular electrical stimulation — quadriceps strenghthening with neuromuscular electrical stimulation (medical device)
  Arms: neuromuscular electrical stimulation
Device: cycle ergometer training — quadriceps strenghthening with cycle ergometer training
  Arms: cycle ergometer training
Other: Conventional pulmonary rehabilitation — excercise training on treadmill

SUMMARY:
The aim of this study is to evaluate the effectiveness of quadriceps strengthening with neuromuscular electrical stimulation versus cycle ergometer as part of pulmonary rehabilitation program , in patients with severe or very severe COPD , according to GOLD with BODE index ≥ 5 .

DETAILED DESCRIPTION:
It's a prospective ,multicentre,randomised, single-blind study which compare the effectiveness of quadriceps strengthening with neuromuscular electrical stimulation versus cycle ergometer training as part of pulmonary rehabilitation program.

The program lasts from 3 to 4 weeks. 102 patients will included, diagnosed with COPD stages GOLD III and IV, and BODE index ≥ 5.

The commun program: training protocol performed on treadmill,quadriceps resistance training,patient therapeutic education,collective gymnastics,relaxation, session psychological care, smoking cessation program and nutritional management if necessary.

The primary criterion is the one minute sit to stand test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD stage 3 or 4, with BODE index ≥ 5
* Hospitalized in the pulmonary rehabilitation unit in the hospital of Morlaix or in the center "Les Acacias" of briançon, with a 3 at 4 weeks pulmonary rehabilitation course;

Exclusion Criteria:

* FEV ≥ 50%
* Pneumonectomy, Lobectomy less than 6 months
* Contraindications to muscle electrostimulation quadriceps
* Absence of written consent
* Inability to follow the respiratory rehabilitation program in its entirety
* People equipped with electronic devices such as pacemakers and intracardiac defibrillators
* Skin lesions and infectious foci on the electrode placement area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
functional capacity of the lower limb muscles | 21 - 4 days / +7 days
  Measure of the functional capacity of the lower limb muscles with the "1 minute Sit To Stand Test "

SECONDARY OUTCOMES:
Maximal isometric voluntary quadriceps strength assessment | 21 - 4 days / +7 days
  Quadriceps strength assessment with handheld dynamometer
isometric voluntary quadriceps endurance assessment | 21 - 4 days / +7 days
  Measure of isometric voluntary quadriceps endurance assessment with handheld dynamometer
assessment of exercise capacity | 21 - 4 days / +7 days
  Six minute walking test for assessing exercise capacity
Quality of Life Assessment | 21 - 4 days / +7 days
  COPD assessment test for assessing quality of life
Dyspnea Assessment with Borg scale | 21 - 4 days / +7 days
  Measure of dyspnea with Borg scale at the end of the six minute walking test
Dyspnea Assessment with MRC Scale | 21 - 4 days / +7 days
  Measure of dyspnea with Medical Research Council Dyspnea Scale
Dyspnea Assessment with Dyspnea 12 questionnary | 21 - 4 days / +7 days
  Measure of dyspnea with Dyspnea 12 questionnary
Inspiratory capacity (in litres) by spirometry | 21 - 4 days / +7 days
  Measure of inspiratory capacity (in litres) by spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Francis Couturaud, MD, PhD, Principal Investigator — University Hospital, Brest
Locations (2):
- France (2):
  - Centre des maladies respiratoires et allergiques - Les Acacias, Briançon, France
  - CH de Morlaix, Morlaix, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Peran L, Beaumont M, Le Ber C, Le Mevel P, Berriet AC, Nowak E, Consigny M, Couturaud F. Effect of neuromuscular electrical stimulation on exercise capacity in patients with severe chronic obstructive pulmonary disease: A randomised controlled trial. Clin Rehabil. 2022 Aug;36(8):1072-1082. doi: 10.1177/02692155221091802. Epub 2022 Apr 11. PMID 35404157
- Available data/document: Clinical Study Report: 22116795 — http://www.ncbi.nlm.nih.gov/pubmed — Vivodtzev I, Debigaré R, Gagnon P, and al. Vivodtzev I, Debigaré R, Gagnon P, Mainguy V, Saey D, Dubé A, Paré MÈ, Bélanger M, Maltais F. Functional and muscular effects of neuromuscular electrical stimulation in patients with severe COPD: a randomized clinical trial. Chest. 2012 Mar;141(3):716-25.
- Available data/document: Clinical Study Report: 24418570 — http://www.ncbi.nlm.nih.gov/pubmed — Vieira PJ, Chiappa AM, Cipriano G Jr, Umpierre D, Arena R, Chiappa GR. Neuromuscular electrical stimulation improves clinical and physiological function in COPD patients.Respir Med. 2014 Apr;108(4):609-20.
- Available data/document: Clinical Study Report: 23440837 — http://www.ncbi.nlm.nih.gov/pubmed — Maddocks M, Gao W, Higginson IJ, Wilcock A.Neuromuscular electrical stimulation for muscle weakness in adults with advanced disease. Cochrane Database Syst Rev. 2013 Jan 31;1.
- Available data/document: Clinical Study Report: 16806873 — http://www.ncbi.nlm.nih.gov/pubmed — Ozalevli S, Ozden A, Itil O, Akkoclu A. Comparison of the Sit-to-Stand Test with 6 min walk test in patients with chronic obstructive pulmonary disease. Respir Med 2007;101(2):286-93.